CLINICAL TRIAL: NCT01443832
Title: Effect of Dephytinisation of Fonio With Intrinsic Wheat Phytase on Iron Absorption in Beninese Women
Brief Title: Iron Absorption From Iron-fortified Fonio Porridge: a Stable Isotope Study
Status: Completed | Type: Observational
Sponsor: Wageningen University (Other)
Collaborators: International Foundation for Science (IFS) (Other)
Responsible Party: Sponsor
Other Study IDs: 10/12 Fonio Study Benin; 005/CNPERS/SA (Other: National Ethical committee (CNPERS-BENIN Republic))
Record Dates: First submitted 2011-09-13; First posted 2011-09-30 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Iron Deficiency
Keywords: ferrous sulfate; iron absorption; Beninese women; fonio
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 2 samples of 8 ml venous blood per subject
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- iron absorption
  Interventions: Dietary Supplement: Fe57 and Fe58-FeSO4 stable isotopes

INTERVENTIONS:
Dietary Supplement: Fe57 and Fe58-FeSO4 stable isotopes — [57Fe] and [58Fe]- FeSO4 prepared from isotopically enriched 57Fe and 58Fe respectively, by dilution of each compound in 0.1 mol H2SO4/L.
  Other Names: iron ferrous sulfate

SUMMARY:
The study sought to investigate the effect of lowering phytic acid in fonio porridge with phytase activity naturally occurring in wheat flour on iron absorption using labelled stable isotopes of iron. The study population is represented by 16 apparently healthy young Beninese women aged 18-30 years recruited based on their willingness to participate and according to inclusion criteria. Test meals consisted of fonio porridges fortified with isotopically labelled [57Fe] or [58Fe] ferrous sulfate with and without wheat flour. Meals were administered to fasting subjects on two consecutive days using a randomised crossover design: half the subjects received the test meal on the first day and the control on the second day and vice versa. Venous blood sample were collected (day 1 and day 14) for iron status and iron absorption measurement. Iron absorption measurement is based on erythrocyte incorporation of iron stable isotope labels 14 days after intake of the labelled test meals and calculated based on isotope-dilution.

DETAILED DESCRIPTION:
Objective: To compare the bioavailability of iron in fonio porridge fortified with isotopically enriched [57Fe] or [58Fe]-ferrous sulfate with and without reducing phytic acid by native phytase in wheat flour.

Study population: Sixteen apparently healthy young women aged 18-30 years recruited at the University based on their willingness to participate and according to inclusion criteria.

Study design: Fonio porridges fortified with isotopically labelled [57Fe] or [58Fe] ferrous sulfate, with (test meal) and without wheat flour (control meal) are administered to fasting subjects on two consecutive days using a randomised crossover design. Half the subjects received the test meal on the first day and the control on the second day and vice versa. No food or drink was allowed within the 3 hours after consumption. All meals were administered under close supervision. Venous blood sample were collected (day 1 and day 16) for iron status and iron absorption measurement. Iron absorption measurement is calculated based on iron isotope-dilution in erythrocyte 14 days after intake of the labelled meals.

Study parameters: Fourteen days before the test, height and weight were measured for nutritional status and subjects were screened for pregnancy and malaria. They were also treated with antihelminth (albendazole tablet). The day before meals test (day 0), whole blood sample was collected for hemoglobin (Hb), serum ferritin (SF), serum Transferrin Receptor (sTfR) and C-reactive protein (CRP). Anemia and iron deficiency was defined as Hb < 120 g/L, and SF < 12 µg/L respectively. Pregnancy test and malaria tests were repeated on that day. On day 1 and day 2, the fonio porridges were randomly given to the subjects on a cross-over designed. Fourteen days after the meal test (day 16) whole blood sample was collected for iron absorption measurement.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 30 y-old
* apparently healthy
* body weight < 65 kg (confirmed by anthropometric measurement at recruitment)
* not pregnant (confirmed by pregnancy test)
* not lactating (confirmed by age of last child if any)
* no reported chronic medical illnesses (diabetes, rheumatism, high blood pressure, etc)
* no reported symptoms of malaria in the last 2 months (fever, headache, stomachache, diarrhoea, nausea, vomiting) (confirmed by malaria test)
* No severe anemia (Hb<90 g/l)
* no intake of vitamin and mineral supplements in the last 2 weeks
* no iron medication or supplementation during the study
* no blood donation in the last 6 months
* no reported allergy to gluten

Exclusion Criteria:

* body weight (> 65 kg)
* pregnant
* recent fever malaria
* abnormal CRP level (>10 mg/l)
* severe anemia (Hb < 90g/l) and iron deficiency (serum ferritin concentration < 12 µg/l)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: apparently healthy young women of reproductive age (18-30y)
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
iron absorption ratio | 14 days
  iron isotopes Fe57 and Fe58 concentration in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Inge D Brouwer, Dr Ir, Study Director — Division of Human Nutrition/Wageningen University
Locations (1):
- Department Nutrition and Food Science/Univsersity of Abomey calavi, Cotonou, Littoral Department, Benin

REFERENCES:
- [Background] Moretti D, Zimmermann MB, Wegmuller R, Walczyk T, Zeder C, Hurrell RF. Iron status and food matrix strongly affect the relative bioavailability of ferric pyrophosphate in humans. Am J Clin Nutr. 2006 Mar;83(3):632-8. doi: 10.1093/ajcn.83.3.632. PMID 16522911